CLINICAL TRIAL: NCT00765401
Title: An Investigation of the Association Between Helicobacter Pylori Infection and Abdominal Pain in Cystic Fibrosis Patients
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: 29239
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cystic Fibrosis; Abdominal Pain; Helicobacter Pylori Infection
Keywords: Abdominal Pain; Cystic Fibrosis; H. pylori; Children
MeSH Terms: conditions — Cystic Fibrosis; Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: The subject with positive breath Test for H.pylori and/or positive stool antigen test
- Group B: The subject with negative breath Test for H.pylori and negative stool antigen test

SUMMARY:
Cystic fibrosis (CF) is the most common lethal autosomal recessive disease among Caucasians. While the pulmonary disease in CF receives most of the attention, gastrointestinal diseases occur in >95% of CF individuals and can contribute to significant morbidity, mortality and a decreased quality of life. The abdominal pain in CF is usual chronic in nature, and the etiology is not usually found, despite medical testing for standard causes of abdominal pain. Helicobacter pylori (Hp) is increasingly being recognized as the etiology of peptic ulcer disease and other upper and lower gastrointestinal tract diseases.1 The role that Hp plays in CF abdominal pain has not been elucidated.

Our long-term goal is to understand relationship between chronic HP infection and abdominal pain in pediatric CF patients.

The specific objective of this proposal is to utilize current state-of-the-art testing for HP to determine the prevalence of Hp in our CF patients age 5 and older.

The central hypothesis is that Cystic fibrosis subjects with significant abdominal pain will have an increased incidence of Helicobacter pylori as determined by the urea breath test and stool antigen test.

The rationale for the proposed research is that once we elucidate a causal relationship between CF patients with abdominal pain and Hp, we can begin treatment of this infection to improve quality of life.

DETAILED DESCRIPTION:
Abdominal pain and Cystic Fibrosis Cystic fibrosis is the most common lethal autosomal recessive disease among Caucasians. CF is caused by a single gene mutation on chromosome 7, which encodes for a membrane protein, the cystic fibrosis transmembrane conductance regulator (CFTR). CFTR channel dysfunction results in progressive pulmonary disease, which is the primary cause of the morbidity and mortality associated with the disease. Therapies directed to slow the progression of the lung disease have increased the USA median survival to 32.2 years.2 Abdominal complaints are very common among CF patients. Littlewood et al. reported that 31% of children had regular complaints of abdominal pain.3 Ravilly et al. performed a retrospective chart review on CF patients referred for treatment to the pain service and those that expired.4 They determined that pain was very common in CF and that 19% of the population had chronic complaints of abdominal pain, which was third behind chest pain and headaches.4 This study likely underestimated the prevalence of abdominal pain in CF, as it was evaluating an end stage lung disease group of patients that were frequently not eating and had severe pain from other disease processes (i.e. headaches from hypercarbia and/or hypoxia, and chest pain from rib fractures).

Known causes of CF related abdominal pain are: 1) malabsorption due to pancreatic steatorrhea, 2) gastroesophageal reflux, 3) esophagitis, 4) gastritis, 5) peptic ulcer disease, 6) pancreatitis, 7) Crohn's disease, 8) distal intestinal obstructive syndrome (DIOS), 9) biliary duct disease including cholocystitis and cholangitis, 10) intussception, 11) acute or chronic gastrointestinal infection, 12) acute appendicitis, and 13) constipation. Given this long list of potential causes, CF patients frequently undergo intensive examinations to determine the etiology of the abdominal pain.4 The testing unfortunately does not always reveal the etiology.

Helicobacter pylori World-wide, Helicobacter pylori (Hp) is increasingly being recognized as the etiology of peptic ulcer disease and other upper and lower gastrointestinal tract diseases.1 With the CF population, The role that Hp plays in abdominal pain has not been elucidated. Two studies have attempted to look at the epidemiology of Hp in CF; however, the approach utilized in those studies was determined to be inadequate. Johansen et al. and Israel et al. both attempted to utilize Hp serology to determine the prevalence in a CF population and determined that there was significant cross-reactivity between Hp and Pseudomonas aeruginosa antigens.10, 11. They concluded that different modes of testing are required if Hp is being evaluated in the CF population. To our knowledge, there have been no further evaluations of Hp in CF using the newer diagnostic tests available.

Testing for Helicobacter pylori Since the isolation of spiral urease-producing Helicobacter pylori bacteria (H. pylori) in 1983 by Drs. Marshall and Warren5, a significant body of evidence has accumulated indicating that the bacteria is an important pathogen in upper GI tract of humans 6,7. The causal relation ship between H.pylori and chronic active gastritis, duodenal ulcer, and gastric ulcer is well documented 8, 9. Methods available for detecting current infection of human stomach by Hp are generally divided into two general types: Invasive and Non-invasive.

Invasive methods include esophageogastroduodenoscopy (EGD) with collection of gastric biopsies. These biopsies are then examined by one or more detection methods: histological examination of stained tissue, microbiological culture of the organism, or direct detection of urease activity in the tissue (for example, the CLO test). Biopsy based methods are expensive, entail greater patient risk and discomfort than non-invasive tests, and may give false negative results due to sampling errors when colonization of the gastric mucosa is patchy 6.

The non-invasive tests include several serological tests that detect serum antibodies to Hp. A positive result with these tests can not distinguish between current infection and past exposure to HP and, therefore, is not a conclusive indicator of current gastrointestinal colonization.

The urea breath test is based on the principal that the urease enzyme is not present in human tissue. Urease presence is indicative of a urease producing organism in the stomach, which is most likely HP. The test has a sensitivity and specificity of 90% and a negative predictive value greater that 95% and a positive predictive value of 90%.12 A third non-invasive test is the Hp stool antigen test also has a sensitivity and specificity of about 90%, and high positive and negative predictive values (>95%).13 Major confounding issues with HP testing are systemic antibiotic exposure, which can lead to false negative tests and partial treatment.14 This is especially problematic in the CF population, who are frequently on systemic antibiotics for chronic suppurative bronchitis. Thus, as part of the inclusion criteria, we will only include subjects who have been off antibiotics for at least 14 days prior to enrollment. The CF patients will be allowed to continue nebulized antibiotics and prophylactic dose of Azythromycin, and analysis will be performed to determine if this results in false negatives by comparing the results to the stool antigen test.

Clinical measures of abdominal pain This study is also designed to determine whether the prevalence of Hp is related to a decreased quality of life, which if documented suggests a pathological role of Hp in CF. Our objective is to use two validated quality of life instruments in this study: The PedsQL (Pediatric Quality of Life Inventory) and the Gastrointestinal Symptom Rating Scale (GSRS).15 The PedsQL is a modular instrument for measuring health-related quality of life (HRQOL) in children and adolescents ages 2 to 18. The PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy-report scales developed as the generic core measure to be integrated with the PedsQL Disease-Specific Modules. The PedsQL 4.0 Generic Core Scales consist of 23 items applicable for healthy school and community populations, as well as pediatric populations with acute and chronic health conditions. The GSRS questionnaire involves 15 items using the Likert scale focusing on gastroesophageal reflux, abdominal pain, constipation, indigestion and diarrhea. It uses a scale from1 to 4.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF by a positive sweat test (more than or equal to 60 mEg/L by quantitative pilocarpine iontophoresis and/ or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with CF phenotype)
2. Abdominal pain during last 6 months
3. Age > 5 and <18 years
4. Either gender

4. Ability to do urea breath test which requires drinking water based solution through a straw and breathing into a breath sample bag 5. Must be off any oral antibiotics and proton pump inhibitors or sucralfate for 14 days.

Subject may continue their prophylactic (X 3/ week) dose of Azithromycin). Patients who are currently on antibiotics or have been on antibiotics within 14 days will be re-screened for inclusion criteria at their next clinic visit (i.e. no wash out).

Exclusion Criteria:

1. Females of child bearing potential with a positive urine pregnancy test The decision not to include pregnant females is based on: 1) the quality of life screens are not designed for pregnancy, 2) their abdominal complaints may be related to pregnancy, 3) safety of the breath test has not been established during pregnancy.
2. Inability to do urea breath test which requires drinking water based solution through a straw and breathing into a breath sample bag.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be enrolled from CF population seen at the Milton S. Hershey Medical Center CF center if they meet the inclusion and exclusion criteria at their scheduled out patient visit to CF clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of Helicobacter pylori in pediatric CF patients. | About a year

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States